CLINICAL TRIAL: NCT05082025
Title: Phase 2 Study of PI3K Inhibitor Copanlisib in Combination With Fulvestrant in Selected ER+ and/or PR+ Cancers With PI3K (PIK3CA, PIK3R1) and/or PTEN Alterations
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Copanlisib development was discontinued by Bayer following withdrawal of copanlisib in relapsed follicular lymphoma in November 2023.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1241; NCI-2021-09936 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2021-09-02; First posted 2021-10-18 (Actual); Results first posted 2025-07-11 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Cancer; Ovarian Cancer
MeSH Terms: conditions — Endometrial Neoplasms; Ovarian Neoplasms | interventions — copanlisib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1: Dose confirmation (Experimental): Up to 6 evaluable patients to confirm a single combination dose of copanlisib and fulvestrant
  Interventions: Drug: Copanlisib; Drug: fulvestrant
- Part 2: Dose expansion: (Experimental): The dose expansion part will enroll in 3 indication-specific cohorts with 13 to 26 patients
  Interventions: Drug: Copanlisib; Drug: fulvestrant

INTERVENTIONS:
Drug: Copanlisib — Given by IV
Drug: fulvestrant — Given by IM

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of copanlisib in combination with fulvestrant in advanced hormone receptor-positive (HR+) solid tumors harboring alterations that activate the Phosphatidylinositol-3 kinase (PI3K) pathway.

DETAILED DESCRIPTION:
Part 1: Dose confirmation:

Primary Objective:

• To evaluate the safety, tolerability, and dose-limiting toxicities (DLT) of copanlisib 60 mg administered intravenously (IV) on Days 1, 8 and 15 in combination with fulvestrant 500 mg administered intramuscularly (IM) on Day 1 and Day 15 of Cycle 1, and then on Day 1 of each subsequent 28-day cycle to confirm the recommended phase 2 doses (RP2D) of the combination therapy.

Secondary objective:

* To assess the efficacy of copanlisib administered in combination with fulvestrant as outlined in Part 2 by evaluating the objective response rate (ORR).
* To evaluate additional efficacy measures such as progression-free survival (PFS) and overall survival (OS) of copanlisib in combination with fulvestrant.

Exploratory Objectives:

• To investigate target engagement, clonal evolution, and mechanisms of resistance using tissue and liquid biopsies utilizing circulating tumor DNA (ctDNA) as outlined in Part 2.

Part 2: Dose expansion:

Primary objectives:

• To assess the efficacy of copanlisib administered in combination with fulvestrant as outlined above by evaluating the objective response rate (ORR). Patients enrolled for Part 1 will be included in this efficacy analysis.

Secondary Objectives:

* To evaluate additional efficacy measures such as PFS and OS of copanlisib in combination with fulvestrant.
* To evaluate the safety and tolerability of copanlisib in combination with fulvestrant.

Exploratory Objectives:

• To investigate target engagement, clonal evolution, and mechanisms of resistance using tissue and liquid biopsies utilizing ctDNA.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed ER+ and/or PR+ advanced or metastatic solid cancer including ovarian cancer (cohort 1), endometrial cancer (cohort 2), or breast cancer (cohort 3) (Figure 1). ER and/or PR positivity is defined as >10% immunohistochemical staining of any intensity. Cohort 3 will be enriched to include at least 7 patients naive to any PI3Ki in Stage 1 and also in Stage 2.
2. Presence of one or more PI3K and/or PTEN alterations in tumor tissue. Genetic alterations will include PIK3CA gain of function mutations, PIK3R1 loss of function mutations, PTEN loss of function mutations, and PTEN deletions.
3. Measurable disease per the RECIST 1.1.
4. The patient (or legally acceptable representative, if applicable) provides written informed consent for the study.
5. Female or male ≥18 years of age on the day of informed consent signing.
6. Patients have no available standard therapy known to prolong survival. For cohort 3 only, prior treatment with aPI3Ki or everolimus is not required and patients with or without prior PI3Ki or everolimus will be qualified for enrollment
7. Adequate archived tumor tissue for the analysis for PI3K and PTEN alterations if available.
8. Eastern Cooperative Oncology Group (ECOG) performance status of .2.
9. Adequate organ and marrow function as defined below:

   1. Hemoglobin ≥ 9.0 g/dL
   2. Absolute neutrophil count ≥1.5 x 10^9/L
   3. Platelet count ≥ 100 x 10^9/L
   4. Total bilirubin (TB) ≤1.5 × institutional upper limit of normal (ULN); Patients with known Gilbert's disease who have TB ≤3 × ULN may be enrolled)
   5. Aspartate transaminase (AST)/ alanine transaminase (ALT) ≤3 × ULN. If patient has liver metastases, AST and ALT ≤5.0 × ULN.
   6. Creatinine ≤1.5 x ULN
   7. International normalized ratio ≤1.5.
10. Fasting blood glucose ≤140 mg/dL and hemoglobin A1c ≤8.5% (both criteria have to be met).
11. Cardiac ejection fraction ≥45%.
12. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 14 days prior to the initiation of treatment and/or postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Women of childbearing potential (WOCBP) must agree and commit to the use of 2 highly effective methods of birth control throughout the duration of the study until at least 150 days following the last dose of study drug. Acceptable methods are defined as those that result, alone or in combination, in a low failure rate (i.e., less than 1% per year) when used consistently and correctly, such as surgical sterilization, an intrauterine device, or hormonal contraception in combination with a barrier method. Women using systemically acting hormonal contraceptives should add a barrier method. In certain countries (if permitted by law), WOCBP may agree to abide by heterosexual sexual abstinence during the time of participation in this study.
13. Male patients and their female partners of childbearing potential must agree and commit to use a barrier contraception (eg, condom with spermicidal foam/gel/film/cream/suppository) throughout the duration of the study until at least 90 days following the last dose of study drug, in addition to their female partners using either an intrauterine device or hormonal contraception and continuing until at least 90 days following the last dose of study drug. This criterion may be waived for male patients who have had a vasectomy > 6 months before signing the ICF.
14. Willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.

Exclusion Criteria:

1. The patient has central nervous system (CNS) involvement. If the patient fulfills the following 3 criteria, she/he is eligible for the study:

   1. Completed prior therapy (including radiation and/or surgery) for CNS metastases, and
   2. CNS tumor is radiologically stable for ≥ 28 days prior to study start, and
   3. The patient is not receiving steroids and enzyme-inducing antiepileptic medications for brain metastases.
2. Patients with HER2 positive breast cancer.
3. Patients must be ≥4 weeks or at least 5 half-lives beyond treatment with any chemotherapy or other investigational therapy including hormonal, biological, or targeted agents at the time of treatment initiation.

   - NOTE: If the patient received major surgery, she/he must have recovered adequately from the toxicity and/or complications from the intervention prior to starting the study treatment.
4. Prior treatment with fulvestrant or any PI3Ki for cohorts 1 and 2.
5. Known hypersensitivity to copanlisib or fulvestrant, or to any of the excipients of copanlisib or fulvestrant.
6. Concomitant use of strong cytochrome P450 (CYP)3A4 inducers (e.g., rifampicin, phenytoin, carbamazepine, phenobarbital, St. John's wort) or inhibitors (e.g., ritonavir, saquinavir, nelfinavir, boceprevir, telaprevir, ketoconazole, omeprazole). Use of strong inhibitors and/or inducers of CYP3A4 is not permitted from Day -14 of Cycle 1 until the start of the study intervention.
7. The patient is currently receiving warfarin or other coumarin derived anticoagulants for treatment, prophylaxis, or otherwise. Therapy with heparin, low molecular weight heparin, fondaparinux, or direct oral anticoagulants such as rivaroxaban or apixaban is allowed.
8. Known additional malignancy that is progressing or requires active treatment.
9. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient fs participation for the full duration of the study or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
10. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
11. Known history of human immunodeficiency virus infection.
12. History or current symptomatic pneumonitis.
13. Has clinically significant, uncontrolled heart disease and/or recent cardiac events, including any of the following:

    1. History of angina pectoris, symptomatic pericarditis, or myocardial infarction within 12 months prior to study entry
    2. History of documented congestive heart failure (New York Heart Association functional classification III-IV)
    3. Documented cardiomyopathy
    4. History of any cardiac arrhythmias, e.g., ventricular, supraventricular, nodal arrhythmias, or conduction abnormality in the previous 12 months
    5. Uncontrolled hypertension defined by a systolic blood pressure (BP) ≥140 mmHg and/or diastolic BP ≥90 mmHg, with or without antihypertensive medication over the course of one clinic visit at intervals of ≥30 minutes. Initiation or adjustment of antihypertensive medication(s) is allowed prior to screening.
14. Type 1 diabetes mellitus.
15. Uncontrolled type 2 diabetes mellitus.
16. Positive cytomegalovirus (CMV) polymerase chain reaction (PCR) test at baseline.
17. Active hepatitis B virus (HBV; chronic or acute; defined as having a known positive hepatitis B surface antigen [HbsAg] test at the time of screening) or hepatitis C infection requiring treatment.

    * Participants with past HBV infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HbcAb] and absence of HbsAg) are eligible if HBV DNA is negative.
    * Participants with positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV RNA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2025-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Yap, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase 2 single center study performed at MD Anderson Cancer Center. Participants were eligible if they had histologically confirmed ER+ and/or PR+ advanced or metastatic ovarian, endometrial, or breast cancers, defined as ≥10% nuclear staining by immunohistochemistry, and confirmed genomic alterations in PIK3CA, PIK3R1, or PTEN.
Pre-assignment Details: Only seven patients were treated on dose level 1 in the Part 1dose confirmation part of the study. The dose expansion phase did not occur.
Groups:
- Part 1: Dose Confirmation - Dose Level 1: Copanlisib 60 mg IV, Days 1, 8, and 15 + Fulvestrant 500 mg IM, Days 1 and 15.
Period: Overall Study
Arm/Group | Part 1: Dose Confirmation - Dose Level 1
Started | 7
Completed | 6
Not Completed | 1
Not completed — Not evaluable for DLT per protocol (dosing less than 1 full cycle of treatment) | 1

BASELINE CHARACTERISTICS:
Population: All 7 patients treated in Part 1: dose confirmation.
Arm/Group | Part 1: Dose Confirmation - Dose Level 1
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 58.7 [34 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT)
Description: A DLT is defined as an intervention-related adverse event that impedes a patient from dosing a full cycle of copanlisib (3 doses), a delay of over 1 week in intitated study intervention occurring secondary to any study related adverse event, or death not clearly attrubuted to an underlying disease or alternate cause. Six out of the seven treated patients were evaluable for DLT. One patient was not evaluable for DLT due to not completing a full cycle of treatment within the first 28-days of treatment.
Time Frame: Within the first cycle (28-days) of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose Confirmation - Dose Level 1
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Number of Participants With Treatment-related Adverse Events
Description: Treatment-related adverse events that were deemed as possibly, probably, or definitely related to treatment, and were graded based on the Common Terminology Criteria for Adverse Events (CTCAE) Version 5. All treatment-related adverse events were captured from the time of signing consent through 30 days after the last dose of study drug or initation of a new anticancer therapy, whichever occurred first. The number of patients experiencing each treatment related adverse event (at least once) is reported.
Time Frame: Through study completion, an average of 14 weeks.
Population: All 7 patients treated in Part 1: dose confirmation.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose Confirmation - Dose Level 1
Number analyzed (Participants) | 7
Participants
  Hyperglycemia | 3
  Fatigue | 3
  Mucositis Oral | 2
  Rash maculo-papular | 3
  Anemia | 1
  Diarrhea | 1
  Nausea | 1
  Pancreatitis | 1
  Flatulence | 1

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 14 weeks
Description: Incidence and causality of all adverse events for all patients treated on-study of all grades and attribution and were graded based on the Common Terminology Criteria for Adverse Events (CTCAE) Version 5. All adverse events were captured from the time of signing consent through 30 days after the last dose of study drug or initiation of a new anticancer therapy, whichever occurred first.
Arm/Group | Part 1: Dose Confirmation - Dose Level 1
All-Cause Mortality (participants affected / at risk) | 4/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Dose Confirmation - Dose Level 1 (N=7)
Back pain (Musculoskeletal and connective tissue disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Dose Confirmation - Dose Level 1 (N=7)
Abdominal pain (Gastrointestinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Anemia (Blood and lymphatic system disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Burn (Skin and subcutaneous tissue disorders) | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 1
cough (Respiratory, thoracic and mediastinal disorders) | 1
creatinine increased (Investigations) | 1
diarrhea (Gastrointestinal disorders) | 2
edema limbs (General disorders) | 2
Fall (General disorders) | 1
Fatigue (General disorders) | 3
Flatulence (Gastrointestinal disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Insomnia (General disorders) | 1
Lymphedema (Vascular disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Neck edema (General disorders) | 1
pain (General disorders) | 1
Pericardian Effusion (Cardiac disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Skin Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT05082025/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT05082025/ICF_001.pdf